CLINICAL TRIAL: NCT06398067
Title: A Pilot Randomized Controlled Trial of Self-Help Plus Stress Management Intervention Among Breast and Gynecologic Cancer Patients in Viet Nam
Brief Title: Stress Management Intervention Among Breast and Gynecologic Cancer Patients in Viet Nam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-44411; K01TW012174 (NIH)
Record Dates: First submitted 2024-04-27; First posted 2024-05-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: Self-Help Plus (SH+); Stress management; Viet Nam; World Health Organization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A 2-arm, parallel, single-blind randomized controlled trial (RCT).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vietnamese Self-Help Plus (vSH+) (Experimental): Participants randomized into this arm will attend information sessions and receive the Vietnamese Self-Help Plus (vSH+) intervention and a copy of the illustrated guide, 'Doing What Matters inn Times of STress' (DWM).
  Interventions: Behavioral: Vietnamese Self-Help Plus (vSH+); Other: 'Doing What Matters in Times of Stress' (DWM) Guide
- Enhanced Usual Care (Active Comparator): Participants randomized into this arm will receive usual care and a copy of the illustrated guide, 'Doing What Matters inn Times of STress' (DWM).
  Interventions: Other: 'Doing What Matters in Times of Stress' (DWM) Guide

INTERVENTIONS:
Behavioral: Vietnamese Self-Help Plus (vSH+) — vSH+ is a stress management program delivered through four 75-minute sessions. It includes the five core SH+ skills. Healthcare workers (nurses and social workers) function as lead facilitators (called 'HW Facilitators') and cancer survivors as co-facilitators (called 'Peer Facilitators').
  Arms: Vietnamese Self-Help Plus (vSH+)
Other: 'Doing What Matters in Times of Stress' (DWM) Guide — An illustrated guide developed by WHO to equip people with practical skills to help cope with stress which has been translated to Vietnamese and reviewed and revised by the investigators.

SUMMARY:
Psychological distress is common among Vietnamese cancer patients but often underestimated and not detected by professionals due to lack of time and overload of clinical work. Currently no established, evidence-based intervention exists to help address the mental health needs of cancer patients in Viet Nam besides the 'Stronger Together' peer mentoring intervention model that the investigators piloted in 2021-2023. The goal of this 2-arm, parallel, single-blind randomized controlled trial (RCT) is to pilot and evaluate the Vietnamese Self Help Plus (vSH+) stress management intervention among breast and gynecologic cancer patients in Viet Nam.

Aim 1- the investigators pilot the adapted vSH+ intervention. After recruitment and screening, participants are randomized into either the intervention (vSH+) or enhanced usual care (EUC) study arms. Participants are invited to attend an in-person informational session (IS) specific to their study arm, where informed consent is obtained.

Aim 2- the investigators assess the potential effectiveness of the vSH+ intervention. Quantitative surveys of study outcomes measures are administered at three timepoints: T0 (baseline, in-person, during info-sessions); T1 (1-2 weeks post-intervention, via phone); and T2 (3 months post-intervention, via phone).

Aim 3- the investigators conduct a qualitative process evaluation, via in-depth interview (IDIs) and focus group discussions (FGDs), to assess the acceptability and feasibility implementing and scaling up the vSH+ intervention model. Satisfaction surveys will be administered during vSH+ sessions and in-depth interviews (IDIs) will be conducted following the conclusion of the intervention. IDIs wil also be conducted with Facilitators, in addition to evaluation surveys during vSH+ sessions and supportive supervision sessions. Between T1 and T2, the investigators will conduct IDIs with Healthcare Workers and focus group discussions with Caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Have a clinician-confirmed diagnosis within the past 12 months of first-time breast and/or gynecologic cancer (e.g., cervical, ovarian, uterine, vaginal, vulvar) in stages I-III
* Currently or will receive treatment with curative intent
* Score less than 8 on the National Comprehensive Cancer Network (NCCN) Distress Thermometer, indicating low to moderate levels of distress
* Score less than 15 on the Patient Health Questionnaire-9 items (PHQ-9, indicating low to moderate levels of depression

Exclusion Criteria:

* Selected '2 Several days' or '3 Almost everyday' on PHQ9 item #9, indicating indicating imminent risk of suicide
* Have severe chronic diseases (e.g., coronary heart disease, chronic obstructive pulmonary disease (COPD), chronic renal failure), at the discretion of the treating clinician or study investigator
* People with a risk for psychosis, mania, and alcohol abuse, based on screening questions commonly used in the field
* Cannot attend the intervention activities at the hospital during the proposed intervention period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in severity of depression | Baseline, 1 month, 3 months
  The Patient Health Questionnaire-9 items (PHQ-9) is a 9 item questionnaire with each item scored from 0 to 3. Scores can range from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Change in Anxiety | Baseline, 1 month, 3 months
  The Generalized Anxiety Disorder-7 items Scale (GAD-7) is a 7 item instrument with each item scored between 0 and 3 where 0=not at all, and 3= nearly every day. Scores can range from 0 to 21 and are interpreted as-- scores 0-4: Minimal Anxiety, scores 5-9: Mild Anxiety, scores 10-14: Moderate Anxiety, and scores greater than 15: Severe Anxiety.

SECONDARY OUTCOMES:
Change in general quality of life | Baseline,1 month, 3 months
  General quality of life will be assessed using the EuroQol 5 Dimensions 5 Levels Questionnaire (EQ-5D-5L). The five dimensions include: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension is rated at five different levels from no problems to the most extreme problems. The questionnaire also includes a visual analog scale asking respondents to rate their current health from 0 (worst health imaginable) to 100 (best health imaginable)
Change in quality of life related to cancer patients' health | Baseline, 1 month, 3 months
  Quality of life related to cancer patients' health will be measured using the Functional Assessment of Cancer Therapy - General, version 4 (FACT-G). This questionnaire includes 27 questions to evaluate 4 domains: physical, social/family, emotional, and functional. Each question is rated on a scale from 0 (not at all) to 4 (very much) based on the patient's experience over the last 7 days.
Change in cancer coping | Baseline, 1 month, 3 months
  Cancer coping will be measured using the Mini-Mental Adjustment to Cancer Scale (Mini-MAC). It consists of five scales: helpless/hopeless, anxious preoccupation, fighting spirit, cognitive avoidance, and fatalism. It has 29 tems on a 4-point Likert scale: 1 (definitely does not apply) to 4 (definitely applies).

OTHER OUTCOMES:
Psychological flexibility (Mediator) | Baseline, 1 month, 3 months
  Mediation analyses will evaluate psychological flexibility, measured by the Acceptance and Action Questionnaire-II (AAQ-2), which is the intended mechanism targeted by SH+. The AAQ2 has 7 items on a 7-point Likert scale: 1 (never true) to 7 (always true).
Social support (moderator) | Baseline, 1 month, 3 months
  Moderation analyses will evaluate social support, assessed with the Medical Outcomes Study Social Support Survey 19 items (MOS-SSS). It assesses four domains of perceived social support: tangible support, emotional-information support, positive social interactions, and affectionate support. Likert response scale range from 1 (none of the time) to 5 (all of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Phuongthao Le, PhD, Principal Investigator — Boston University
Locations (6):
- Vietnam (6):
  - Can Tho Oncology Hospital, Can Tho
  - Oncology Center, Cho Ray Hospital, Chợ Rây
  - Da Nang Oncology Hospital, Da Nang
  - Breast and Gynecology Department, Hung Vuong Women's Hospital, Ho Chi Minh City
  - Ho Chi Minh City Oncology Hospital, Ho Chi Minh City
  - Oncology Center, Hue Central Hospital, Huế

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le PD, Nguyen NB, Dang ATT, Tran LTK, Pham HN, Le TA, Vo KV, Nguyen HT, Hoang DT, Phan DC, Nguyen CBT, Nguyen MHT, Nguyen QH, Phan HNT, Dang TQ, Nguyen HT, Le DD, Phan THT, Nguyen PTN, Nguyen VT, Tran PT, Pham AN, Vom Eigen K, Campbell R, Taylor C, Tran HTT, Hoang MV. Pilot randomised controlled trial of the self-help plus stress management intervention among patients with breast and gynaecological cancer in Viet Nam: a study protocol. BMJ Open. 2025 Dec 17;15(12):e106185. doi: 10.1136/bmjopen-2025-106185. PMID 41407411